CLINICAL TRIAL: NCT05370001
Title: Does Endotracheal Tube (ETT) Size Facilitate Carbon Dioxide Washout in Liver Tumour Ablation With High Frequency Jet Ventilation (HFJV)? - a Randomised Controlled Trial
Brief Title: Endotracheal Tube Size Effect on the Carbon Dioxide Washout During Jet Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ETT-size Karolina Galmén
Record Dates: First submitted 2022-04-25; First posted 2022-05-11 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-05

CONDITIONS: Liver Tumor
Keywords: high frequency jet ventilation; endotracheal tube size; carbon dioxide; liver tumor ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Patients planned for liver tumour ablation will be randomised to one of two sizes of ETT, size 8 or size 9.
Who Masked: Participant
Masking Description: The patient is not being informed what ETT-size is being used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine procedure - use of ETT size 9 (No Intervention): When using HFJV in liver tumour ablation procedures for optimizing surgical conditions, an ETT size 9 is routinely being used in our department.
- Experimental group - use of ETT size 8 (Experimental): In this arm an endotracheal tube of size 8 will be used. This is one size smaller than is routine when HFJV is being used for liver tumour ablation procedures in our department. Worth to note is that an endotracheal tube of size 8 is routine in all other surgical procedures, in men, during general anaesthesia.
  Interventions: Other: Entotracheal tube size

INTERVENTIONS:
Other: Entotracheal tube size — Compare the levels of carbon dioxide and if it is related to ETT size when using size 9 (routine) or size 8 (intervention).
  Arms: Experimental group - use of ETT size 8

SUMMARY:
High Frequency Jet Ventilation (HFJV) can be used in liver tumour ablation to minimise breathing related movements. The jet cannula is placed freely inside an endotracheal tube (ETT) and the outflow of air is passive, moving out in the interspace between the jet cannula and the inner walls of the ETT.

This study aims to investigate whether the tube size can influence the washout of carbon dioxide using two different sizes of ETT's.

DETAILED DESCRIPTION:
The aim of the present prospective randomised study is to compare differences in levels of carbon dioxide between two different endotracheal tube-sizes.

Background: High Frequency Jet Ventilation (HFJV) has become an important technique for ventilation during stereotactic near-diaphragm ablation to minimise breathing related movements. Thus, avoiding risks associated to movements and subsequent dislocation of the target tumour. HFJV is being increasingly used during CT-guided, percutaneous liver tumour ablation. As shown previously, breathing related movements in upper abdominal organs, are decreased significantly when compared to conventional ventilation. When HFJV is being used in the setting for tumour ablation the jet cannula is inserted into an ordinary endotracheal tube (ETT). The HFJV catheter is placed in the ETT and is during jet ventilation lying freely within the tube. Right placement is confirmed by a harmonic curve on the screen of the jet ventilator. It is of great importance that the ETT is not obstructed as this type of ventilation is dependent on passive outflow of expired air, through the tube, passing from the lungs around the catheter within the tube into the surrounding air. If the lumen around the catheter within the ETT is becoming too small, there is a risk for intrinsic PEEP built up, and subsequent risk for barotrauma, pneumothorax. The space between the catheter and the inner lumen of the ETT also governs the exhalation of gas, the passage of expired gas containing CO2 from the lung. A small inner diameter of the ETT may thus likewise increase the risk for a raise in arterial carbon dioxide. To minimise these risks, an ETT one size larger than usual can be used to lower the risk for pressure increase and improve gas exchange. One should consider the risks, even though very low, of mechanical injury in the airway when larger ETT's are being used. Previous studies on arterial blood gas in liver tumour was performed using a ETT one size larger (size 9 in men). Tadié et al showed that laryngeal injury was related to the length of intubation, the non-use of muscle relaxant drugs and the height/ETT diameter ratio. This was a study made in an ICU and all patients were intubated >24 hrs and therefore not fully applicable to the OR-setting. Jaensson et al describe a significant lower risk for post operative sore throat (POST) using a smaller ETT size in women during elective surgery. Myles et al describe women being 1.5 times more likely to report having POST compared to men. To defend the superiority of a larger tube size further studies assessing the effect of the ETT size on the arterial CO2 tension is needed.

Methods: After written, informed consent, 26 (13 in each group) consecutive, male patients planned for liver tumour ablation with HFJV will be included in the study.

Participants will be randomized to ETT size 8 or 9. Randomisation will take place in an earlier stage with the help of a computerised randomisation generator where 26 envelopes are prepared in which the information of tube size is to be found. The envelopes are on the outside anonymous. The envelopes will be opened by the anaesthetic nurse in the operation room, who will then prepare the ETT.

An arterial line will be placed before the start of anaesthesia and a transcutaneous measuring device will be placed on the forehead of the patient. After preoxygenation, induction and ETT placement, conventional ventilation will be started and a normal tcCO2 value reached (tcCO2 4,5-5 before the start of HFJV). HFJV will have pre-set settings with the same values for all patients. Driving pressure (DP) will be 1,2 bar and frequency 220/min. Measurements from the three different methods; arterial pCO2, transcutaneous CO2 and etCO2 will then be recorded at the start of HFJV (t=0) and then every 15' until t=45 minutes of HFJV. In the case of rapidly increasing CO2, a cut off limit of 10 kPa will be used. When this level is reached, settings on the ventilator will be changed. That means increasing DP and, if needed, lower the frequency. If this does not lead to a satisfactory CO2-level HFJV has to be changed to conventional ventilation until the CO2-level is within normal limits. Any injury during intubation and post extubation stridor (PES) will be recorded. The patient will be asked for post operative sore throat (POST) and any signs of postoperative hoarseness (PH) will be noted in the protocol before leaving the post anaesthetic care unit (PACU) and also approximately 24 hrs after extubation. If symptoms still occur after 24 hrs, follow up will take place approximately 72 hrs and 96 hrs after extubation. If symptoms are still present by this point the patient will be offered a doctor's appointment.

Statistics: The power calculation was based on data from previous studies. The base-line PaCO2 among 12 male patients, at the start of HFJV, was 4.9 kPa (SD 0.5) with an increase to mean PaCO2 of 6.7 (SD 1.5) at 15 minutes with HFJV and a tube size of 9. With the hypothesis that the PaCO2 would increase to a mean of 8.0 kPa after 15 minutes of HFJV ventilation, with a tube size 8, groups of 11 patients are needed to verify the difference at a p<0.05 with a power of 80%. To compensate for potential drop-outs, groups of 13 patients is set as the study population. Data will be presented as mean, SD, median and range where applicable. One-way ANOVA will be used on normal distributed data and ANOVA on ranks will be used on non-normal distributed data. Bonferroni's test will be used to compare differences between the different timepoints. A p-value of <0,05 will be considered as statistically significant.

Importance of the study: This study is conducted to if the larger endotracheal tube size has benefits in gas exchange when HFJV is being used in liver tumour ablation procedures. Normally it is desirable to use as small ETT as possible as this minimises the risks for airway injury. The risks of air entrapment and even pneumothorax and raise in carbon dioxide levels are also risks that are potentially harmful for the patients and must be avoided. The small risk of using a one size larger ETT would therefore be accepted if the benefits can be shown in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients scheduled for stereotactic liver tumour ablation.
* Need for an arterial line for safe monitoring of hemodynamic and respiratory variables during the procedure/anaesthesia.
* Ability to understand the information about the study and be able to leave a written, informed consent.

Exclusion Criteria:

* Patients with known CO2 retention.
* Patients shorter than 160 cm (as an endotracheal tube size 9 would then be too big).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As men and women routinely uses two different ETT sizes and we wanted to compare two sizes within one group, this study will only focus on men.
Enrollment: 26 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Carbon dioxide level from an arterial line (PaCO2) after 15 minutes of HFJV. | 15 minutes after the start of HFJV
  Carbon dioxide level from an arterial line (PaCO2) in kPa will be compared from the levels at baseline to the level at 15 minutes of HFJV.

SECONDARY OUTCOMES:
Dynamics of carbon dioxide during surgery using HFJV | From the start of HFJV up until 45 minutes after the start of HFJV
  The dynamics of carbon dioxide changes obtained from an arterial line (PaCO2) in kPa, transcutaneously (tcCO2) in kPa and end tidal measurement (etCO2) in kPa registered every 15 minutes during the first 45 minutes of HFJV. That is, all values from each timepoint (15 minutes, 30 minutes and 45 minutes after the start of HFJV) will be compared to baseline.
During HFJV measure pause pressure (PP) and peak pressure . | From the start of HFJV up until 45 minutes after the start of HFJV
  During HFJV measure pause pressure (PP) in mbar and peak pressure in mbar .
Analysing PaO2 | From the start of HFJV up until 45 minutes after the start of HFJV
  PaO2 in kPa will also be measured and analysed during the procedure.
Analysing pH | From the start of HFJV up until 45 minutes after the start of HFJV
  pH will also be measured and analysed during the procedure.
Analysing lactate | From the start of HFJV up until 45 minutes after the start of HFJV
  Lactate in mmol/L will also be measured and analysed during the procedure.
Analysing saturation | From the start of HFJV up until 45 minutes after the start of HFJV
  Saturation in percent will also be measured and analysed during the procedure.
Injury of the airway following endotracheal intubation. | At the most 96 hours post extubation.
  Signs of apparent mechanical injury in the airway. Signs of apparent injury, being visible injury during intubation and post extubation stridor (PES). Post operative sore throat (POST) and any signs of postoperative hoarseness (PH)

CONTACTS AND LOCATIONS:
Overall Officials: Klara Bergmark, MD, Study Director — Region Stockholm
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung DY, Tse DM, Boardman P, Gleeson FV, Little MW, Scott SH, Anderson EM. High-frequency jet ventilation under general anesthesia facilitates CT-guided lung tumor thermal ablation compared with normal respiration under conscious analgesic sedation. J Vasc Interv Radiol. 2014 Sep;25(9):1463-9. doi: 10.1016/j.jvir.2014.02.026. Epub 2014 May 10. PMID 24819833
- [Background] Denys A, Lachenal Y, Duran R, Chollet-Rivier M, Bize P. Use of high-frequency jet ventilation for percutaneous tumor ablation. Cardiovasc Intervent Radiol. 2014 Feb;37(1):140-6. doi: 10.1007/s00270-013-0620-4. Epub 2013 May 2. PMID 23636246
- [Background] Biro P, Spahn DR, Pfammatter T. High-frequency jet ventilation for minimizing breathing-related liver motion during percutaneous radiofrequency ablation of multiple hepatic tumours. Br J Anaesth. 2009 May;102(5):650-3. doi: 10.1093/bja/aep051. Epub 2009 Apr 3. PMID 19346232
- [Background] Engstrand J, Toporek G, Harbut P, Jonas E, Nilsson H, Freedman J. Stereotactic CT-Guided Percutaneous Microwave Ablation of Liver Tumors With the Use of High-Frequency Jet Ventilation: An Accuracy and Procedural Safety Study. AJR Am J Roentgenol. 2017 Jan;208(1):193-200. doi: 10.2214/AJR.15.15803. Epub 2016 Oct 20. PMID 27762601
- [Background] Galmen K, Harbut P, Freedman J, Jakobsson JG. High frequency jet ventilation for motion management during ablation procedures, a narrative review. Acta Anaesthesiol Scand. 2017 Oct;61(9):1066-1074. doi: 10.1111/aas.12950. Epub 2017 Aug 13. PMID 28804874
- [Background] Galmen K, Jakobsson JG, Freedman J, Harbut P. High Frequency Jet Ventilation during stereotactic ablation of liver tumours: an observational study on blood gas analysis as a measure of lung function during general anaesthesia. F1000Res. 2019 Apr 5;8:386. doi: 10.12688/f1000research.18369.1. eCollection 2019. PMID 31583085
- [Background] Tadie JM, Behm E, Lecuyer L, Benhmamed R, Hans S, Brasnu D, Diehl JL, Fagon JY, Guerot E. Post-intubation laryngeal injuries and extubation failure: a fiberoptic endoscopic study. Intensive Care Med. 2010 Jun;36(6):991-8. doi: 10.1007/s00134-010-1847-z. Epub 2010 Mar 18. PMID 20237758
- [Background] Jaensson M, Olowsson LL, Nilsson U. Endotracheal tube size and sore throat following surgery: a randomized-controlled study. Acta Anaesthesiol Scand. 2010 Feb;54(2):147-53. doi: 10.1111/j.1399-6576.2009.02166.x. Epub 2009 Nov 23. PMID 19930246
- [Background] Myles PS, Hunt JO, Moloney JT. Postoperative 'minor' complications. Comparison between men and women. Anaesthesia. 1997 Apr;52(4):300-6. doi: 10.1111/j.1365-2044.1997.89-az0091.x. PMID 9135179